CLINICAL TRIAL: NCT01093573
Title: A Phase I/II Study of Midostaurin (PKC412) and 5-Azacitidine for Elderly Patients With Acute Myelogenous Leukemia.
Brief Title: Midostaurin and Azacitidine in Treating Elderly Patients With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brenda Cooper, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Brenda Cooper, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CASE1908; NCI-2009-01285 (Other: NCI/CTRP)
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Untreated Adult Acute Myeloid Leukemia
Keywords: Untreated myelodysplastic syndromes
MeSH Terms: interventions — midostaurin; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 1 (Experimental): Aza at 75 mg/m2 D1-7 & Midostaurin 25 mg BID D 8-21
  Interventions: Drug: midostaurin; Drug: azacitidine; Other: bone marrow aspiration; Other: mutation analysis; Other: Pharmacokinetic study
- Dose Level 2 (Experimental): Aza at 75 mg/m2 D1-7 & Midostaurin 50 mg BID D 8-21
  Interventions: Drug: midostaurin; Drug: azacitidine; Other: bone marrow aspiration; Other: mutation analysis; Other: Pharmacokinetic study
- Dose Level 3 (Experimental): Azacitidine 75 mg/m2 IV D1-7 & Midostaurin 75 mg PO BID D 8-21
  Interventions: Drug: midostaurin; Drug: azacitidine; Other: bone marrow aspiration; Other: mutation analysis; Other: Pharmacokinetic study

INTERVENTIONS:
Drug: midostaurin — Given orally
  Other Names: N-benzoyl-staurosporine; PKC412
Drug: azacitidine — Given IV
  Other Names: 5-AC; 5-azacytidine; 5-AZC; azacytidine; ladakamycin; Vidaza
Other: bone marrow aspiration — Correlative study: Pretreatment bone marrow aspirates or blood [(3 ml in EDTA tube (purple top)] will be analyzed according to local institution guidelines to determine whether blasts contain wild type Flt3, ITD, or Flt 3 mutations.
Other: mutation analysis — Correlative study
Other: Pharmacokinetic study — Correlative study: Concentrations of unchanged midostaurin and its major metabolites, CGP52421 and CGP62221 in plasma samples will be determined using a validated liquid chromatography / mass spectrometry method.
  Other Names: Pharmacokinetic studies

SUMMARY:
RATIONALE: Midostaurin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Midostaurin may help azacitidine kill more cancer cells by making the cancer cells more sensitive to the drug. PURPOSE: This phase I/II trial is studying the side effects and best dose of midostaurin when given together with azacitidine and to see how well it works in treating elderly patients with acute myelogenous leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safe and tolerable dose of midostaurin in combination with azacitidine in patients with acute myelogenous leukemia. (Phase I) II. To describe the toxicity profile of the combination of midostaurin and azacitidine in patients with acute myelogenous leukemia. (Phase I/II) III. To determine the complete and partial response rate and rate of hematologic improvement of midostaurin and 5-azacitidine in untreated acute myelogenous leukemia. (Phase I/II)

SECONDARY OBJECTIVES:

I. To describe pharmacokinetics of oral midostaurin given in combination with azacitidine on a day 8-21 schedule. (Phase I/II) II. To correlate treatment response with FLT3 mutational status in a descriptive fashion. (Phase I/II) III. To assess overall survival of patients from initiation of midostaurin-azacitidine toxicities. (Phase I/II) IV. To determine median disease-free survival of the regimen in untreated patients. (Phase II)

TERTIARY OBJECTIVES:

I. To describe signaling in CD117+ committed myeloid precursors in whole blood and bone marrow samples before and during treatment. (Phase I/II) II. To measure in vivo FLT3 inhibition using plasma inhibition assay (PIA) and Flt ligand (FL) levels in patients enrolled on this trial before and during treatment. (Phase I/II)

OUTLINE: This is a phase I, dose escalation study of midostaurin followed by a phase II study.

Patients receive azacitidine intravenously (IV) over 10-20 minutes on days 1-7 and midostaurin orally (PO) twice daily (BID) on days 8-21. Courses repeat every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologic proof of active AML at time of enrollment
* Phase I and II portion: Subjects of any age with untreated AML, if not candidates for standard induction chemotherapy or with poor risk AML (i.e. preceding MDS, myeloproliferative syndromes, leukemia due to cytotoxic chemotherapy for another condition, adverse cytogenetics or complex karyotype), or any subjects > 70 years of age with untreated AML. Acute promyelocytic leukemia (FAB M3) is excluded
* Please note: prior intensive induction therapy for acute leukemia is allowed only in the phase I portion of this study

  • PHASE I PORTION ONLY: Patients of any age who have received no more than one prior attempt at induction chemotherapy (and may have received treatment consolidation), must have recovered from acute toxicities of therapy and be >= 4 weeks from last dose of cytotoxic treatment; patients who have received prior autologous or allogeneic stem cell transplantation are not eligible; patients may have received 1 or 2 cycles of cytarabine-based therapy as attempted induction.
* Phase II portion: Patients must have not received any prior intensive induction therapy for AML.

  * Intensive induction includes standard induction chemotherapy such as 7 & 3, high dose cytarabine, mitoxantrone-etoposide, low-dose subcutaneous cytarabine.
  * Allowed "non-intensive" prior treatments for pre-existing hematologic conditions (i.e., MDS, chronic myelomonocytic leukemia [CMML]) will include: hydroxyurea, thalidomide, hematopoietic growth factors, Zarnestra, Lenalidomide, arsenic, Imatinib, and corticosteroids, suberoylanilide hydroxamic acid [SAHA] inhibitors; hydroxyurea is allowed up to 24 hours before initiating treatment and to control blood counts during the first cycle of chemotherapy after azacitidine has completed; a minimum of 4 weeks must have elapsed since the administration of thalidomide, Zarnestra, Revlimid, arsenic, SAHA inhibitors, or any investigational medication; a minimum of five days must have elapsed since the administration of growth factors

    * Prior cytotoxic chemotherapy for another condition treated with curative intent is allowed provided at least 18 months has elapsed between last treatment and enrollment on protocol
    * Eastern Cooperative Oncology Group (ECOG) performance status 0-2
    * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 1.5 times the upper limits of normal
    * Serum bilirubin =< 1.5x upper limit of normal
    * Creatinine =< 1.5x upper limit of normal
    * No exclusion for blood counts; however, at the time of treatment initiation, white blood cell (WBC) should be < 30,000/uL (can be controlled with hydroxyurea)
    * Life expectancy without treatment of at least 12 weeks
    * Patients with and without FLT3 mutations will be eligible to participate
    * Patients must have the ability and willingness to sign a written informed consent document

Exclusion Criteria

* Acute promyelocytic leukemia (FAB M3)
* Prior autologous or allogeneic stem cell transplant
* Prior azacitidine, decitabine, or midostaurin
* Patients with known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of midostaurin; patients with gastric bypass surgery are excluded
* Patients with any other known active cancer (except carcinoma in-situ), concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, pulmonary, chronic renal disease, active uncontrolled infection)
* Cardiovascular Criteria will exclude a patient from participation in the study will include:

  * Screening electrocardiogram (ECG) with a QTc > 450 msec;
  * Patients with congenital long QT syndrome;
  * History or presence of sustained ventricular tachycardia;
  * Any history of ventricular fibrillation or torsades de pointes;
  * Bradycardia defined as heart rate (HR) < 50 bpm;
  * Right bundle branch block + left anterior hemiblock (bifascicular block);
  * Patients with myocardial infarction or unstable angina < 6 months prior to starting study drug;
  * Congestive heart failure (CHF) New York (NY) Heart Association class III or IV;
  * Patients with an ejection fraction =< 45% assessed by multi gated acquisition scan (MUGA) or echocardiogram (ECHO) scan within 14 days of day 1
  * Poorly controlled hypertension
* Known allergy or hypersensitivity to azacitidine, mannitol, or midostaurin
* Active or suspicion of central nervous system (CNS) leukemia
* Patients with human immunodeficiency virus (HIV) disease or active viral hepatitis
* Patients with hepatitis B
* Patients with an abnormal chest X-ray and/or any pulmonary infiltrate including those suspected to be of infectious origin; in particular, patients with resolution of clinical symptoms of pulmonary infection but with residual pulmonary infiltrates on chest x-ray are not eligible until pulmonary infiltrates have completely resolved
* Pregnant or lactating women
* Prohibited medications: PKC412 and its two major metabolites may have a potential of drug-drug interactions with P-gp substrates and CYP3A4 inhibitors, and inducers. An increased anticoagulant effect has been noted in patients treated with warfarin and midostaurin.
* Patients who have received any investigational agent within 30 days prior to day 1
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months of midostaurin medication. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
  * Combination of any two of the following (a+b or a+c, or b+c):

    1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment Sexually active males unless they use a condom during intercourse while taking drug and for 5 months after stopping midostaurin medication. They should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-07; Primary Completion 2016-09-08 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Cooper, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Background] Tomlinson BK, Gallogly MM, Kane DM, Metheny L, Lazarus HM, William BM, Craig MD, Levis MJ, Cooper BW. A Phase II Study of Midostaurin and 5-Azacitidine for Untreated Elderly and Unfit Patients With FLT3 Wild-type Acute Myelogenous Leukemia. Clin Lymphoma Myeloma Leuk. 2020 Apr;20(4):226-233.e1. doi: 10.1016/j.clml.2019.10.018. Epub 2019 Nov 6. PMID 32085993

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Aza at 75 mg/m2 D1-7 & Midostaurin 25 mg BID D 8-21
  midostaurin: Given orally
  azacitidine: Given IV
  bone marrow aspiration
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 3 | 3 | 28
Completed | 3 | 3 | 26
Not Completed | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Insurance Denied | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 3 | 3 | 28 | 34
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 0 | 0 | 1 | 1
  60-69 years | 1 | 1 | 4 | 6
  70-79 years | 1 | 2 | 16 | 19
  80-89 years | 1 | 0 | 7 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 15 | 19
  Male | 1 | 1 | 13 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 28 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 4 | 5
  White | 3 | 2 | 24 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 28 | 34

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Midostaurin in Combination With Azacitidine in Patients With Acute Myelogenous Leukemia (Phase I)
Description: Patients received azacitidine 75 mg/m intravenous over 30 minutes daily for 7 consecutive days followed by escalating doses of oral midostaurin (25 mg bid, 50 mg bid, and 75 mg bid) days 8-21. Determination of the maximum tolerated dose (MTD) was based on dose-limiting toxicities (DLT) observed during the first cycle of treatment
Time Frame: Day 28
Population: All participants who received treatment for the Phase I part of the study
Measure: Number; unit: mg/bid
Groups:
- Midostaurin Dose Escalation: Patients receive Azacitidine at 75 mg/m2 D1-7 & Midostaurin (25 mg bid, 50 mg bid, and 75 mg bid) mg BID D 8-21
  midostaurin: Given orally
  azacitidine: Given IV
Arm/Group | Midostaurin Dose Escalation
Number analyzed (Participants) | 11
mg/bid | 75

2. Primary Outcome: Number of Participants With Hematologic Improvement (Phase I)
Description: Number of participants with HI. Hematologic improvement (HI): must last at least 2 months in the absence of ongoing cytotoxic therapy and will be another endpoint of interest (although it will not be considered in the final statistical analysis) and will be defined according to IWG criteria .
Time Frame: After 2 cycles of therapy
Population: Participants that received treatment on the phase I portion of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Patients receive azacitidine at 75 mg/m2 D1-7 & Midostaurin 25 mg BID D 8-21
  midostaurin: Given orally
  azacitidine: Given IV
  .
- Dose Level 2: Patients receive azacitidine at 75 mg/m2 D1-7 & Midostaurin 50 mg BID D 8-21
- Dose Level 3: Patients receive azacitidine at 75 mg/m2 D1-7 & Midostaurin 75mg BID D 8-21
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 3 | 3 | 11
Participants | 0 | 0 | 2

3. Primary Outcome: Overall Response Rate (Phase II)
Description: Number of participants with CR, CRi, PR and Hematologic improvement (HI). Response will be assessed using the standard morphologic criteria for acute leukemia as follows: Complete remission (CR): ANC ≥ 1000/ uL and platelets of > 100,000/ uL without circulating blasts and bone marrow with < 5% blasts and no Auer rods; Morphologic complete remission with incomplete blood recovery (CRi): Patients fulfills all of the criteria for remission except for residual neutropenia (ANC < 1000/ uL) or thrombocytopenia (platelet count < 100,000/uL). Partial remission (PR): This designation requires at least a 50% decrease in the bone marrow blasts to 5-25%.
Time Frame: after 4 months of treatment
Population: All participants that received at least 2 cycles of treatment at the MTD (Dose Level 3)
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 3: Patients receive azacitidine at 75 mg/m2 D1-7 & Midostaurin 75 mg BID D 8-21
  midostaurin: Given orally
  azacitidine: Given IV
Arm/Group | Dose Level 3
Number analyzed (Participants) | 24
Participants
  Complete Remission (CR) | 4
  Complete Remission with incomplete recovery (CRi) | 1
  Partial Remission | 2
  No remission/response | 17
  Hematologic improvement without CR/PR | 0

4. Primary Outcome: Toxicity Profile (Phase II)
Description: Number of patients experiencing at least one instance of specific treatment emergent adverse events
Time Frame: during treatment up to 10 cycles
Population: Participants that received at least one dose of midostaurin at the MTD (Dose Level 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 3
Number analyzed (Participants) | 24
Participants | 24

5. Secondary Outcome: Duration of Response
Description: Time to progression after confirmed response
Time Frame: Up to 3 years
Population: All participants on phase II (dose level 3) that were evaluable for response.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Level 3
Number analyzed (Participants) | 7
days | 252 [14 to 517]

6. Secondary Outcome: Overall Survival (Phase II)
Description: Median time of overall survival of participants from initiation of midostaurin-azacitidine
Time Frame: Up to 3 years
Population: All participants that received treatment at the MTD (dose level 3)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Level 3
Number analyzed (Participants) | 24
days | 244 [203 to 467]

7. Secondary Outcome: Correlate Treatment Response With FLT3 Mutational Status in a Descriptive Fashion.(Phase I)
Description: Number of participants with FLT3 mutation that had a response to treatment
Time Frame: Baseline to 4 cycles (16 weeks)
Population: There were no subjects with FLT3 mutation, there for this outcome measure has no data.
Groups:
- Azacitidine and Midostaurin: Patients receive azacitidine IV over 10-20 minutes on days 1-7 and oral midostaurin twice daily on days 8-21.
  midostaurin: Given orally
  azacitidine: Given IV
  bone marrow aspiration: Correlative study: Pretreatment bone marrow aspirates or blood [(3 ml in EDTA tube (purple top)] will be analyzed according to local institution guidelines to determine whether blasts contain wild type Flt3, ITD, or Flt 3 mutations.
  mutation analysis: Correlative study
  Pharmacokinetic study: Correlative study: Concentrations of unchanged midostaurin and its major metabolites, CGP52421 and CGP62221 in plasma samples will be determined using a validated liquid chromatography / mass spectrometry method.
Arm/Group | Azacitidine and Midostaurin
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Pharmacokinetic Profile of Midostaurin Given With Azacitidine (Phase I)
Description: Change in Midostaurin trough levels and active metabolite levels between cycles one and two
Time Frame: after 2 cycles
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes of Phosphorylation Status of FLT3 in Blood and Bone Marrow Samples (Phase I/II)
Time Frame: Baseline to 4 cycles (16 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events collected while participants were on study for up to 3 years.
Groups:
- Dose Level 1; Dose Level 2; Dose Level 3: Patients receive azacitidine IV over 10-20 minutes on days 1-7 and oral midostaurin twice daily on days 8-21.
  midostaurin: Given orally
  azacitidine: Given IV
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 3/28
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 22/28
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=28)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1/26 (1)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 6 (6)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis-2ndary to AML (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=28)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (7) | 4 (5)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 3 (19) | 2 (42) | 19 (138)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 2 (4) | 12 (25)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
bilateral lower extremity lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 3 (7)
Bloody nose (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Boil: right axilla (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (5)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (5) | 2 (4) | 15 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 9 (11)
Creatinine increased (Investigations) | 2 (3) | 0 (0) | 12 (34)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
diaphoretic (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 2 (3) | 15 (22)
Dizziness (Nervous system disorders) | 1 (3) | 1 (1) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 12 (22)
E. Petechiae infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ecchymoses: skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (3) | 0 (0) | 10 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 4 (4)
erythemia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (8) | 2 (5) | 15 (51)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Fever (General disorders) | 2 (2) | 1 (1) | 5 (8)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 6 (10)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
hemorrhage-right eye (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (4)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 3 (12) | 14 (37)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6) | 3 (10) | 5 (17)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 13 (23)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 1 (5) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 2 (7) | 1 (5) | 9 (28)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 7 (8)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection w/grade 3 ANC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection: parotoditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Inflammation: picc site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (11)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
left axilla mass (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
left leg/leukemia cutis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
lesion on foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lightheadedness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (6) | 3 (25) | 10 (75)
Mucositis oral (Gastrointestinal disorders) | 1 (3) | 0 (0) | 6 (10)
Muffled hearing (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3) | 15 (26)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (7) | 3 (31) | 16 (82)
Non-blood (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
occassional night sweats (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5)
Pain (General disorders) | 1 (2) | 1 (1) | 8 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 5 (6)
Patorid swelling-right (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Peeling skin/fingerprints (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (5)
Penile infection-abcess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 4 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PICC Line Inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (21) | 3 (52) | 22 (160)
Pneumonia-probable fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Rash- knees and back (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Renal burning (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Right hand infection, cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Shingles reactivation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Skin break down buttocks-abcess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Stuffy nose (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
subconjuctival hemorrhage right eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (3) | 11 (18)
Weight loss (Investigations) | 0 (0) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (4) | 2 (39) | 11 (88)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes